CLINICAL TRIAL: NCT05582304
Title: Role of Glare and Spectral Filtering on Contrast Sensitivity: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6501
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- TEST/CONTROL/Photopic CSF (Experimental): Eligible subjects who are habitual wearers of silicone hydrogel contact lenses will be randomized to the photopic condition and randomized contralaterally to the TEST/CONTROL lenses.
  Interventions: Device: Test Lens; Device: Control Lens
- TEST/CONTROL/Mesopic CSF (Experimental): Eligible subjects who are habitual wearers of silicone hydrogel contact lenses will be randomized to the mesopic condition and randomized contralaterally to the TEST/CONTROL lenses.
  Interventions: Device: Test Lens; Device: Control Lens
- CONTROL/TEST/Photopic CSF (Experimental): Eligible subjects who are habitual wearers of silicone hydrogel contact lenses will be randomized to the photopic condition and randomized contralaterally to the CONTROL/TEST lenses.
  Interventions: Device: Test Lens; Device: Control Lens
- CONTROL/TEST/Mesopic CSF (Experimental): Eligible subjects who are habitual wearers of silicone hydrogel contact lenses will be randomized to the mesopic condition and randomized contralaterally to the CONTROL/TEST lenses.
  Interventions: Device: Test Lens; Device: Control Lens

INTERVENTIONS:
Device: Test Lens — ACUVUE OASYS MAX 1-Day with TearStable Technology and OptiBlue Light Filter
Device: Control Lens — ACUVUE OASYS 1-Day with HydraLuxe Technology

SUMMARY:
This will be a split-plot design, randomized, parallel, double-masked feasibility study to evaluate the role of a test lens on contrast sensitivity with and without glare.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 65 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear spherical silicone hydrogel soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
5. Possess a wearable pair of spectacles that provide correction for distance vision.
6. The spherical equivalent of the subject's vertex corrected distance refraction must be between -1.00 D and -6.00 D (inclusive) in each eye.
7. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be between 0.00 D and 1.00 D (inclusive) in each eye.
8. The best corrected, monocular, distance visual acuity must be 20/25 or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Be currently pregnant or lactating.
2. Be currently using any ocular medications or have any ocular infection of any type.
3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
5. Be currently wearing monovision or multifocal contact lenses.
6. Be currently wearing lenses in an extended wear modality.
7. Have participated in a contact lens or lens care product clinical trial within 30 days prior to study enrollment.
8. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site.
9. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
10. Have a history of strabismus or amblyopia.
11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
12. Have had any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).
13. Have signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar).
14. Have a history of eyelid injury, surgery or procedure that resulted in abnormal eyelid position or movement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a split-plot design with two parallel arms consisting of two randomized lighting conditions (photopic and mesopic). Within each parallel arm, subjects were further randomized in a contralateral fashion to the Test and Control lenses. A total of 40 subjects were enrolled and completed the study.
Groups:
- Photopic: OD: Test (Senofilcon A C3) / OS: Control (Senofilcon A C3): Subjects randomized to this condition arm and lens sequence received the Test lens on the right eye and received the Control lens on the left eye under the photopic condition.
- Photopic: OD: Control (Senofilcon A C3) / OS: Test (Senofilcon A C3): Subjects randomized to this condition arm and lens sequence received the Control lens on the right eye and received the Test lens on the left eye under the photopic condition.
- Mesopic: OD: Test (Senofilcon A C3) / OS: Control (Senofilcon A C3): Subjects randomized to this condition arm and lens sequence received the Test lens on the right eye and received the Control lens on the left eye under the mesopic condition.
- Mesopic: OD: Control (Senofilcon A C3) / OS: Test (Senofilcon A C3): Subjects randomized to this condition arm and lens sequence received the Control lens on the right eye and received the Test lens on the left eye under the mesopic condition
Period: Overall Study
Arm/Group | Photopic: OD: Test (Senofilcon A C3) / OS: Control (Senofilcon A C3) | Photopic: OD: Control (Senofilcon A C3) / OS: Test (Senofilcon A C3) | Mesopic: OD: Test (Senofilcon A C3) / OS: Control (Senofilcon A C3) | Mesopic: OD: Control (Senofilcon A C3) / OS: Test (Senofilcon A C3)
Started | 9 | 11 | 11 | 9
Completed | 9 | 11 | 11 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects administered a study lens.
Groups:
- Photopic: Subjects assigned bright light conditions (~120 cd/m2).
- Mesopic: Subjects assigned dim light conditions (~3cd/m2).
- Total: Total of all reporting groups
Arm/Group | Photopic | Mesopic | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (14.14) | 37.1 (13.95) | 37.4 (13.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 4 | 2 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 2 | 3
  Black or African American | 1 | 2 | 3
  White | 18 | 16 | 34
Region of Enrollment [Number; unit: Participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Photopic Contrast Sensitivity Function Under Bright Light Conditions (∼120 cd/m2) With a Broadband Glare Source
Description: Photopic contrast sensitivity was measured under bright light conditions (~120 cd/m2) with a broadband glare source at five spatial frequencies (1.6, 3.2, 8, 16 and 24 cpd) using the University of Georgia system. The area under the log contrast sensitivity function (AULCSF) was derived by first calculating the logarithm of contrast sensitivity as logCS = log10(contrast sensitivity), and then AULCSF was calculated using logCS and the log (base 10) of each spatial frequency based on the trapezoidal rule per eye per subject. The AULCSF was computed by trapezoidal integration of the logarithm of the contrast sensitivity (vertical axis) as a function of the logarithm of spatial frequency (horizontal axis). The unit of the horizontal axis is log(cpd) since spatial frequency is in the unit of cycles per degree (cpd). Although, sensitivity is a unitless parameter, to aid interpretation, the units of AULCSF are described as log(sensitivity)*log(cpd).
Time Frame: Up to 2 hours post-fitting
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: log(sensitivity)*log(cpd)
Units Other Than Participants: eyes
Groups:
- Test (Senofilcon A C3): Subject eyes that wore the Test lens during the study.
- Control (Senofilcon A C3): Subject eyes that wore the Control lens during the study.
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 20 | 20
log(sensitivity)*log(cpd) | 1.92 (0.220) | 1.62 (0.158)

2. Secondary Outcome: Area Under the Curve of Mesopic Contrast Sensitivity Under Dim Light Conditions (∼3 cd/m2) With a Broadband Glare Source.
Description: Mesopic contrast sensitivity was measured under dim light conditions (~3 cd/m2) with a broadband glare source at five spatial frequencies (1.6, 3.2, 8, 16 and 24 cpd) using the University of Georgia system. The area under the log contrast sensitivity function (AULCSF) was derived by first calculating the logarithm of contrast sensitivity as logCS = log10(contrast sensitivity), and then AULCSF was calculated using logCS and the log (base 10) of each spatial frequency based on the trapezoidal rule per eye per subject. The AULCSF was computed by trapezoidal integration of the logarithm of the contrast sensitivity (vertical axis) as a function of the logarithm of spatial frequency (horizontal axis). The unit of the horizontal axis is log(cpd) since spatial frequency is in the unit of cycles per degree (cpd). Although, sensitivity is a unitless parameter, to aid interpretation, the units of AULCSF are described as log(sensitivity)*log(cpd).
Time Frame: Up to 2 hours post-fitting
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol.
Measure: Mean (Standard Deviation); unit: log(sensitivity)*log(cpd)
Units Other Than Participants: eyes
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 20 | 20
log(sensitivity)*log(cpd) | 0.57 (0.189) | 0.43 (0.140)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately three hours per subject.
Groups:
- Test (Senofilcon A C3): Subjects that wore the Test lens in either eye during the study.
- Control (Senofilcon A C3): Subjects that wore the Control lens in either eye during the study.
Arm/Group | Test (Senofilcon A C3) | Control (Senofilcon A C3)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT05582304/Prot_SAP_000.pdf